CLINICAL TRIAL: NCT07389148
Title: Evaluation of Salivary Cortisol Levels and Physiological Stress Parameters in Children With Molar Incisor Hypomineralization: A Comparative Observational Study
Brief Title: Salivary Cortisol Levels in Children With Molar Incisor Hypomineralization
Status: Recruiting | Type: Observational
Sponsor: Lokman Hekim University (Other Government)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Hamide Comert, Assistant Professor, Specialist in Pediatric Dentistry, Lokman Hekim University
Other Study IDs: 2025054
Record Dates: First submitted 2026-01-22; First posted 2026-02-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Molar incisor hypomineralization; Salivary cortisol; Dental anxiety; Physiological stress; Children; Pediatric dentistry
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples collected using an absorption-based method for cortisol analysis. Samples will not be used for genetic testing or DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MIH Group: Children aged 8 to 12 years diagnosed with molar incisor hypomineralization (MIH) according to the European Academy of Paediatric Dentistry (EAPD) criteria. Participants in this group undergo a routine clinical dental examination without any therapeutic intervention. Physiological stress parameters, including salivary cortisol levels, heart rate, and oxygen saturation, are assessed during the dental visit.
- Control Group: Age- and sex-matched healthy children aged 8 to 12 years without a diagnosis of molar incisor hypomineralization. Participants undergo a routine clinical dental examination without any therapeutic intervention. Salivary cortisol levels, heart rate, and oxygen saturation are measured using the same protocol as applied to the MIH group.

SUMMARY:
Molar incisor hypomineralization (MIH) is a developmental condition that affects the enamel of permanent molars and incisors in children and may cause tooth sensitivity, discomfort, and difficulties during dental treatment. These problems can increase dental anxiety and lead to physiological stress responses during dental visits.

The purpose of this observational study is to evaluate physiological stress responses in children with MIH by measuring salivary cortisol levels, heart rate, and oxygen saturation, and to compare these findings with those of children without MIH. A total of 90 children aged 8 to 12 years will participate in the study, including 45 children diagnosed with MIH and 45 healthy control participants.

Participation involves no treatment or intervention beyond a routine clinical dental examination. Heart rate and oxygen saturation will be measured during the dental visit, and saliva samples will be collected immediately after the examination using a non-invasive method to assess cortisol levels. The results of this study may contribute to a better understanding of stress responses in children with MIH and support the development of more individualized and anxiety-sensitive dental care approaches.

DETAILED DESCRIPTION:
Molar incisor hypomineralization (MIH) is a developmental enamel defect that may lead to hypersensitivity, discomfort during dental procedures, and increased dental anxiety in affected children. While behavioral aspects of anxiety in children with MIH have been investigated, objective assessment of physiological stress responses in this population remains limited.

This prospective observational study is designed to evaluate physiological stress responses in children with MIH by assessing salivary cortisol levels in conjunction with non-invasive physiological parameters recorded during a routine dental examination. The study includes a comparative design involving children with an MIH diagnosis and healthy control participants.

All procedures are conducted under standardized clinical conditions to minimize external factors that may influence stress responses. Saliva samples are collected using a non-invasive absorption-based method immediately after the dental examination to assess cortisol levels. Physiological parameters are recorded at predefined time points during the dental visit to capture stress-related changes associated with the clinical environment.

The study aims to provide objective data on stress-related physiological responses in children with MIH, which may contribute to improved understanding of anxiety-related mechanisms and support the development of more individualized, child-centered dental care strategies.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 8 and 12 years.
* Children diagnosed with molar incisor hypomineralization (MIH) according to the European Academy of Paediatric Dentistry (EAPD) criteria or healthy children without MIH.
* Ability to cooperate sufficiently to complete the clinical dental examination and study procedures.
* Written informed consent obtained from a parent or legal guardian.

Exclusion Criteria:

* Presence of systemic, hormonal, or metabolic diseases.
* Regular use of medications known to affect salivary cortisol levels or cardiovascular parameters (e.g., corticosteroids, beta-blockers).
* History of systemic conditions that may influence stress response.
* Refusal of participation by the child or parent/legal guardian.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consists of children aged 8 to 12 years attending the Department of Pediatric Dentistry. Participants include children diagnosed with molar incisor hypomineralization and age-matched healthy control children without MIH.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-04-26 (Estimated)

PRIMARY OUTCOMES:
Salivary Cortisol Level | Day 1 (Immediately after the clinical dental examination)
  Salivary cortisol concentration measured immediately after the routine clinical dental examination as an objective biomarker of physiological stress.

SECONDARY OUTCOMES:
Heart Rate | Day 1 (During the clinical dental examination)
  Heart rate measured using a pulse oximeter during the routine clinical dental examination to assess physiological stress response.
Oxygen Saturation (SpO₂) | Day 1 (During the clinical dental examination)
  Peripheral oxygen saturation measured using a pulse oximeter during the routine clinical dental examination as a physiological parameter associated with stress response.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Faculty of Dentistry, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the pediatric nature of the study and ethical considerations regarding participant confidentiality.

REFERENCES:
- [Background] Schwendicke F, Elhennawy K, Reda S, Bekes K, Manton DJ, Krois J. Global burden of molar incisor hypomineralization. J Dent. 2018 Jan;68:10-18. doi: 10.1016/j.jdent.2017.12.002. Epub 2017 Dec 6. PMID 29221956
- [Background] Weerheijm KL, Duggal M, Mejare I, Papagiannoulis L, Koch G, Martens LC, Hallonsten AL. Judgement criteria for molar incisor hypomineralisation (MIH) in epidemiologic studies: a summary of the European meeting on MIH held in Athens, 2003. Eur J Paediatr Dent. 2003 Sep;4(3):110-3. PMID 14529329
- [Background] Jalevik B, Sabel N, Robertson A. Can molar incisor hypomineralization cause dental fear and anxiety or influence the oral health-related quality of life in children and adolescents?-a systematic review. Eur Arch Paediatr Dent. 2022 Feb;23(1):65-78. doi: 10.1007/s40368-021-00631-4. Epub 2021 Jun 10. PMID 34110616
- [Background] Contac LR, Pop SI, Dobreanu M, Oprica M, Voidazan S, Bica CI. Salivary Cortisol as a Biomarker for Assessing Fear and Anxiety in Patients with Molar-Incisor Hypomineralization. Diagnostics (Basel). 2025 Feb 17;15(4):489. doi: 10.3390/diagnostics15040489. PMID 40002640